CLINICAL TRIAL: NCT07203235
Title: Investigations of The Relationship Between Core Function Aand Endurance, Gait Speed, Balance, and Proprioception in Transtibial Amputees
Brief Title: The Investigations of Core Muscles, Gait, Balance and Proprioception in Transtibial Amputees
Status: Completed | Type: Observational
Sponsor: sevilay seda bas (Other)
Responsible Party: Sponsor-Investigator, sevilay seda bas, Asst. Prof., Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: 08/932
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amputee Group: This group consists of individuals aged between 18 and 50 years who have undergone a unilateral transtibial amputation and have been using a prosthesis for at least 6 months. Participants must have a Medicare Functional Classification Level (MFCL) of K2 or higher, indicating the ability to ambulate in the community. Individuals with neurological or mental disorders, recent (past 12 months) orthopedic problems other than amputation, pregnancy, or those who use walking aids will be excluded.
  Interventions: Other: evaluation
- Control Group: This group includes healthy individuals aged between 18 and 50 years with no history of amputation. Participants must not have any neurological or mental disorders, recent orthopedic issues (within the past 12 months), or pregnancy, and must not use walking aids.
  Interventions: Other: evaluation

INTERVENTIONS:
Other: evaluation — Participants will undergo a series of evaluations including core muscle function tests, endurance assessments, proprioceptive measurements, balance testing, and gait analysis. These assessments are non-invasive and observational, aimed at comparing functional performance between individuals with transtibial amputation and healthy controls. No interventions will be applied; only assessments will be conducted.

SUMMARY:
The goal of this observational study is to investigate the effects of transtibial amputation on core function and endurance, and their relationship with proprioception, balance, and gait in adults with transtibial amputation and healthy controls.

The main questions it aims to answer are:

Do individuals with transtibial amputation show reduced core function and endurance compared to non-amputees?

Is there a relationship between core function/endurance and proprioception, balance, and gait performance in transtibial amputees?

Researchers will compare individuals with transtibial amputation to non-amputee individuals to see if there are significant differences in core endurance, posture, and functional abilities.

Participants will:

Perform tests to assess core function and muscular endurance

Undergo evaluations of proprioception, balance, and gait

ELIGIBILITY:
Inclusion Criteria (for Amputee Group):

* Age between 18 and 50 years
* Unilateral transtibial amputation
* Use of a prosthesis for at least 6 months
* Medicare Functional Classification Level (MFCL) of K2 or higher (indicating the ability to ambulate in the community)
* Willingness to participate and provide informed consent

Inclusion Criteria (for Control Group):

* Age between 18 and 50 years
* Willingness to participate and provide informed consent

Exclusion Criteria (for Amputee Group):

* Presence of any neurological disorder
* Presence of any mental health disorder
* Any orthopedic condition (other than amputation) within the past 12 months
* Pregnancy
* Use of a walking aid (e.g., cane, walker)

Exclusion Criteria (for Control Group):

* Presence of any neurological disorder
* Presence of any mental health disorder
* Any orthopedic condition within the past 12 months
* Pregnancy
* Use of a walking aid (e.g., cane, walker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will be conducted at Ankara Yıldırım Beyazıt University and at private prosthetics and orthotics centers in Ankara, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Knee Joint Position Sense (Proprioception) | Single assessment at time of participant enrollment
  Position sense of the knee joints in both amputated and intact limbs will be measured using a dual digital inclinometer (ACUMAR™, Lafayette, USA). Participants are instructed and trained before testing. The participant was asked to lie prone with the knee positioned at 40 degrees. After learning this angle, the participant was asked to reproduce the remembered angle independently. The difference between the target angle and the reproduced angle was recorded. This procedure was repeated three times.

SECONDARY OUTCOMES:
Trunk Position Sense (Proprioception) | Single assessment at time of participant enrollment
  Position sense of the trunk will be measured using a dual digital inclinometer (ACUMAR™, Lafayette, USA). Tests are conducted barefoot on a firm surface with eyes closed. Participants are instructed and trained before testing. For trunk position sense, inclinometers are placed on T1 and S1 spinous processes, and participants perform 30-degree trunk flexion movements and then return to neutral, attempting to replicate the angle three times.
Core Muscle Function | Single assessment at time of participant enrollment
  Core muscle function will be assessed by measuring transversus abdominis (TrA) muscle strength using the Stabilizer Pressure Biofeedback Unit (Chattanooga Group Inc, USA). Participants lie prone with pressure set at 70 mmHg and perform the abdominal drawing-in maneuver three times for 10 seconds each; the average pressure change is recorded.
Core Muscle Endurance (Trunk Flexor) | Single assessment at time of participant enrollment
  Core muscle endurance will be evaluated through McGill's endurance tests including trunk flexor, trunk extensor, and lateral plank tests. The trunk flexor test involves maintaining a 55-degree flexion position until the participant can no longer hold it. For all tests, participants will be asked to maintain the position for as long as possible, and the duration will be recorded.
Core Muscle Endurance (Trunk Extansor) | Single assessment at time of participant enrollment
  Core muscle endurance will be evaluated through McGill's endurance tests including trunk flexor, trunk extensor, and lateral plank tests. The trunk extensor test is performed prone with pelvis, hips, and knees stabilized; participants hold a horizontal position until failure. For all tests, participants will be asked to maintain the position for as long as possible, and the duration will be recorded.
Core Muscle Endurance (Lateral Plank) | Single assessment at time of participant enrollment
  Core muscle endurance will be evaluated through McGill's endurance tests including trunk flexor, trunk extensor, and lateral plank tests. The lateral plank test requires participants to maintain a side-lying plank position with the body aligned until loss of form or contact with the ground. For all tests, participants will be asked to maintain the position for as long as possible, and the duration will be recorded.
Balance | Single assessment at time of participant enrollment
  Static balance will be evaluated using the single-leg stance test. Participants are asked to stand unsupported on one leg while maintaining balance. The duration they can hold this position is measured with a stopwatch and recorded in seconds
Gait Speed | Single assessment at time of participant enrollment
  Gait speed will be assessed using the 10-meter walk test. Participants start from a standing position and walk 10 meters at their comfortable walking speed. The time to complete the 10 meters is measured with a stopwatch.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)